CLINICAL TRIAL: NCT06830382
Title: A Multicentre, Prospective, Open-label Study With [68Ga]Ga-ABY-025 PET-imaging to Characterize HER2-expression and Explore the Therapy-predictive Value for HER2-antibody Drug Conjugates in Patients With Metastatic Breast Cancer
Brief Title: HER2-PET as a Precision Imaging Tool for Treatment With HER2-ADC in HER2-expressing mBC
Status: Recruiting | Type: Observational
Sponsor: Renske Altena (Other)
Collaborators: Karolinska Institutet (Other); Affibody (Industry)
Responsible Party: Sponsor-Investigator, Renske Altena, Study Director, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Other Study IDs: HER2-Ex PET; 2024-512721-89-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Stage IV; HER2-low Breast Cancer; Molecular Imaging
Keywords: HER2-PET; molecular imaging; precision imaging; HER2-low mBC; metastatic breast cancer; HER2-ADC; ABY-025
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples for extracellular vesicles; tumor biopsies for proteomics analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm 1: HER2-expressing cohort: Patients are allocated to arm 1 based on HER2-status in the tumor biopsy. Patients in arm 1 are treated - according to approved indications and the current standard of care - with trastuzumab deruxtecan. Patients in arm 1 will undergo a second PET after 3-4 treatment courses (9-12 weeks) and and optional third HER2-PET + tumor biopsy at the moment of disease progression.
  Interventions: Diagnostic Test: Positron emission tomografy with [68Ga]Ga-ABY-025
- Arm 2: HER2-zero cohort: Patients with HER2-zero tumors (according to tumor biopsy) will be followed for possible AE's after the experimental investigation (HER2-PET) during two weeks after the investigation, and will thereafter go off study.
  Interventions: Diagnostic Test: Positron emission tomografy with [68Ga]Ga-ABY-025

INTERVENTIONS:
Diagnostic Test: Positron emission tomografy with [68Ga]Ga-ABY-025 — Investigational Medicinal product (IMP):[68Ga]Ga-ABY-025 (all patients)

SUMMARY:
This is a prospective, multi-center, open-label, exploratory diagnostic phase II imaging trial for patients with metastatic breast cancer with at least one line of systemic therapy.

The overarching aim of the HER2-Ex PET trial is to study the role of precision imaging utilizing positron emission tomography (PET) with the HER2-specific tracer [68Ga]Ga-ABY-025 (hereafter referred to as HER2-PET) in enhancing treatment planning for patients with metastatic HER2-expressing breast cancer Patients will be allocated based on HER2-status on PET and biopsy. Patients with HER2-expressing lesions in a fresh or archived tumour biopsy will be treated with T-DXd.

The study hypothesis is that PET/CT precision imaging with a contemporary HER2-radiotracer ([68Ga]Ga-ABY-025) can be used and can lead to a potentially better identification of patients who benefit from T-DXd treatment, thereby achieving improved treatment responses as well as fewer side effects. This study's diagnostic approach provides a more individualized treatment strategy. Additionally, this study can potentially give us a better biological understanding of HER2-expressing mBC.

DETAILED DESCRIPTION:
The target population of the trial consists of female patients with mBC with known non-HER2-positive tumours or with unknown HER2-status. Patients can be included in the trial at the time of disease progression after at least one line of chemotherapy in the palliative setting, or within six months after completion of adjuvant therapy for primary breast cancer.

Patients will be recruited at the Breast Clinics of the Karolinska Comprehensive Cancer Center in Stockholm, the Uppsala Academic Hospital in Uppsala, and Skåne University hospital in Sweden. Additional study sites may be added during the conduct of the trial and after approval of the regulatory agencies. Patients can be referred for study-related investigations from other sites, but all study-related investigations will be performed at one of the three above-mentioned clinics.

Participants are eligible to participate in the study if they meet all the inclusion and none of the exclusion criteria listed below. Subject eligibility (that participants fulfil all inclusion criteria and do not meet any exclusion criteria) is established by the principal investigator or co- investigator that is involved in clinical care for the patient.

When an eligible patient decides to participate in the study, all screening- and treatment related procedures will be initiated no earlier than after the informed consent form is signed.

All patients will undergo a baseline study-specific HER2-PET and a tumour biopsy, the latter guided by the results from the HER2-PET. Lesions with sonographically feasible access and preferably with ABY-025 tracer uptake SUVmax ≥ 6 will be eligible for biopsy. In case no ABY-025 lesions are present or accessible for biopsy, a non-avid metastatic lesion is recommended for biopsy. For practical reasons, biopsies taken prior to the HER2-PET (no more than three months old and without exposition to systemic anti-cancer therapy or local radiotherapy to the specific lesion) can be used for study purpose.

Patients with HER2-expressing fresh or archived tumour biopsy will be treated with T-DXd.

A second HER2-PET will be done in all patients treated with T-DXd at the moment of treatment response evaluation after 9-12 weeks of treatment with T-DXd. An optional third HER2-PET and tumor biopsy will be done at the moment of disease progression on T-DXd.

ELIGIBILITY:
Inclusion Criteria:

* Female patients age ≥18 years.
* Metastatic or locally advanced breast cancer with disease progression after ≥ 1 line of chemotherapy in the palliative setting, or with disease relapse within six months after completion of (neo-) adjuvant chemotherapy.
* The patient must be able and willing to provide written consent to participate in the study.
* At least one metastatic lesion ≥ 10 mm is available for biopsy

  o Exception can be made when a recent biopsy is available (no more than 12 months old and without exposition to HER2-targeted therapy or local radiotherapy to the specific lesion).
* At least one additional metastatic index lesion ≥ 10 mm for evaluation of treatment effect (according to RECIST v1.1)
* WHO performance status ≤ 2.
* Expected survival > 12 weeks.
* Contraceptives: Females of child-bearing potential must agree to use adequate contraception prior to study entry, for the duration of the study treatment phase and for six months after the last dose of [68Ga]Ga-ABY-025. Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, established, proper use of hormonal contraceptives that inhibit ovulation, hormone- releasing intrauterine devices (IUDs), and copper IUDs. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception. Women must refrain from donating eggs during this same period. Should a female become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately. If a female participant is of child-bearing potential (females are considered not of childbearing potential if they are at least one year postmenopausal and/or surgically sterile), she must have a documented negative serum Pregnancy testing prior to each administration of the IMP is obligatory.

Exclusion Criteria:

* Contra-indications for treatment for trastuzumab deruxtecan and inability to undergo this treatment as per local treatment routines.
* A previously documented metastatic tumor biopsy that was HER2-positive (IHC 3+ and/or HER2 gene amplification).
* Other manifest malignancies except for basal cell carcinoma of the skin.
* Inadequate cardiac, renal, bone marrow or liver function
* Patients with increased risk of complications from biopsies, i.e. increased risk of bleeding, defined as

  * prothrombin time test (INR value) >1.4, platelet count <70 (109/l), activated partial thromboplastin time (APTT) >30s.
  * known bleeding disorders such as haemophilia, von Willebrand disease or platelet disorders.
  * any anticoagulants or antiplatelet treatment that cannot be temporarily paused

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mBC considered for treatment with T-DXd.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2030-04-01 (Estimated); Study Completion 2032-04-01 (Estimated)

PRIMARY OUTCOMES:
Therapy-predictive role of HER2-PET for the clinical benefit of treatment with T-DXd in patients with HER2-expressing mBC | 9-12 weeks (first response evaluation)
  The primary endpoint is the correlation between the mean [68Ga ]Ga-ABY-025 SUVmax in the five most ABY-025 avid lesions at the baseline HER2-PET and treatment response according to RECIST v1.1 after three-four cycles of treatment with T-DXd.

SECONDARY OUTCOMES:
Changes in HER2-status according to [68Ga]Ga-ABY-025 uptake prior to and after 3-4 cycles of treatment with T-DXd | 9-12 weeks (first response evaluation)
  Changes (deltaSUVmax) in HER2-status in up to five target lesions according to [68Ga ]Ga-ABY-025 uptake prior to and after 3-4 cycles of treatment with T-DXd.
Correlation between the proportion of HER2-avid metastases in relation to the total burden of disease (lesions ≥10 mm) on CT and treatment response. | 12 months
  Correlation between HER2-expressing total tumor volume (HER2-TTV; defined as proportion of ABY-025 avid lesions in relation to the total tumor volume (TTV, lesions ≥10 mm) defined on CT) at baseline and Overall Response Rate.
Health related quality of life at baseline, the first response evaluation and at disease progression. | 9-12 weeks (first response evaluation)
  Change in patient reported Health-Related Quality of Life (HR-QoL) as measured by the EQ-5D-5L questionnaire from baseline to the first treatment evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Renske Altena, MD PhD, Study Director — Karolinska Institutet
Locations (1):
- Karolinska University hospital, Solna, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared upon a reasonable request to the study sponsor representative and study director.